CLINICAL TRIAL: NCT03612726
Title: The Overall Survival of Patients Diagnosed With Unresectable Hepatocellular Carcinoma Under Real-life Clinical Practice in Asia Pacific Region
Brief Title: The Overall Survival of Patients With Unresectable HCC in Real-life
Status: Recruiting | Type: Observational
Sponsor: Humanity & Health Medical Group Limited (Other)
Collaborators: Tokyo University (Other)
Responsible Party: Sponsor
Other Study IDs: APASL_HCC_2018V1
Record Dates: First submitted 2018-07-17; First posted 2018-08-02 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Liver cancer is the fifth most common cancer and the second most frequent cause of cancer-related death globally. Hepatocellular carcinoma represents about 90% of primary liver cancers and constitutes a major global health problem. The pattern of HCC occurrence shows a significant geographical imbalance, with the highest incidence rates in East Asia (more than 50% of the cases occurring in China).

The aim of this study is to investigate the overall survival (OS) of patients diagnosed with unresectable hepatocellular carcinoma under real-world practice conditions in Asia Pacific region.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of unresectable hepatocellular carcinoma
* Able to comprehend and provide written informed consent in accordance with institutional guidelines.

Exclusion Criteria:

* Patients not willing to participate and/or give their written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Unresectable HCC who are treated under real-life clinical practice conditions in Asian Pacific Region
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2018-07-16 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | Up to 5 years
  Overall survival (OS) is defined as the time (days) from the date of unresectable HCC diagnosis to the date of death, due to any reason. Patients alive or lost to follow-up at the time of analysis will be censored at their last date of follow-up

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to 5 years
  Progression-free survival (PFS) is defined as the time (days) from the start of treatment to the date of first observed disease progression (radiological or clinical, whichever is earlier) or death due to any cause, if death occurs before progression is documented
Time to progression (TTP) | Up to 5 years
  Time to progression (TTP) is defined as the time (days) from the start of treatment to the first documented disease progression
Duration of treatment | Up to 5 years
  Duration of treatment, defined by the time interval from the start of treatment to the day of permanent discontinuation of treatment (including death)
Frequency and Severity of Adverse Events | Up to 5 years
  Safety will be evaluated by monitoring and recording the grade 3, 4 and 5 adverse events (AE) occurring during and after treatment throughout follow up of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Masao Omata, PhD, MD, Study Chair — Tokyo University; George Lau, MD, Study Chair — Humanity & Health Medical Group Limited
Locations (3):
- Beijing 302 Hospital, Beijing, China
- Humanity & Health Medical Group Limited, Hong Kong, Hong Kong
- Tokyo University, Tokyo, Japan